CLINICAL TRIAL: NCT01339858
Title: The Effect of N-Acetyl Cysteine on Cortical Erosion in Early Stage Schizophrenia
Acronym: Breier-Stanley
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Alan Breier, Psychiatrist, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1008-12
Record Dates: First submitted 2011-04-19; First posted 2011-04-21 (Estimated); Results first posted 2019-05-08 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-04

CONDITIONS: Schizophrenia; Psychotic Disorder NOS; Schizoaffective Disorder; Schizophreniform
MeSH Terms: conditions — Schizophrenia; Mental Disorders; Psychotic Disorders | interventions — Acetylcysteine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N-Acetyl Cysteine (Experimental): NAC and matched placebo will be supplied in unmarked capsules. Each NAC capsule will contain 600 mg of NAC. Dosing will begin at 600 mg/d and titrated up over 5 weeks until a maximum dose of 3600 mg/d is reached. This approximate dose was effective and well tolerated in a recent study of treatment refractory obsessive-compulsive disorder by Krystal and colleagues at Yale (16). In addition, a double-blind placebo controlled trial recently completed at IUSM Riley Hospital in children (age 4 to 12 years) with autism spectrum disorders used doses ranging from 900 mg/day to 4200 mg/day and reported no serious adverse events and found the agent well tolerated (15). Dose adjustments downward to 1920 mg/d will be permitted if tolerability issues are encountered at the maximum dose.
  Interventions: Drug: N-Acetyl Cysteine
- Sugar Pill (Placebo Comparator): matched placebo
  Interventions: Other: sugar pill

INTERVENTIONS:
Drug: N-Acetyl Cysteine — NAC and matched placebo will be supplied in unmarked capsules. Each NAC capsule will contain 480 mg of NAC. Dosing will begin at 480 mg/d and titrated up by 480 mg/d each week until a maximum dose of 2880 mg/d (BID) is reached. This approximate dose was effective and well tolerated in a recent study of treatment refractory obsessive-compulsive disorder by Krystal and colleagues at Yale (16). In addition, a double-blind placebo controlled trial recently completed at IUSM Riley Hospital in children (age 4 to 12 years) with autism spectrum disorders used doses ranging from 900 mg/day to 4200 mg/day and reported no serious adverse events and found the agent well tolerated (15). Dose adjustments downward to 1920 mg/d will be permitted if tolerability issues are encountered at the maximum dose
  Arms: N-Acetyl Cysteine
Other: sugar pill — matched placebo will be supplied in unmarked capsules. Dosing regimen will be the same as in the N-Acetyl Cysteine arm.
  Arms: Sugar Pill

SUMMARY:
The primary objective of this study is to determine if NAC, added to existing antipsychotic treatment, is superior to placebo for cortical erosion in patients with early stage psychosis. The primary hypothesis is that there will be significantly less cortical erosion as measured by cortical thickness, cortical volume and cortical white matter density (assessed by DTI) in patients treated for 12 months with NAC as compared to those treated with placebo. The secondary objectives of this study are to determine if 12 months of NAC add-on treatment is superior to placebo for fMRI determined working memory and semantic memory tasks, cortical MR spectroscopy measures (glutathione, N-acetylaspartate, and glutamine/glutamate levels), electrophysiologically determined attention measures (e.g., mismatch negativity, P300), symptoms, functional measures and cognitive functioning.

DETAILED DESCRIPTION:
Schizophrenia is a severe, debilitating illness that typically begins during the teen-age years and early twenties, and worsens over time as it evolves into a chronic, life-long disorder. Existing treatments suppress psychotic symptoms but do not prevent the evolution of underlying disease processes that results in poor, long term outcomes. Recent studies have shown that progressive erosion of cortical mass occurs during the early stages of schizophrenia (1-3). The investigators hypothesize that arresting cortical erosion during the early phases of schizophrenia will prevent subsequent clinical deterioration and the descending course of illness associated with this disorder. The investigators propose to establish a research program that will assess the ability of agents with neuroprotective properties to halt cortical loss and thereby prevent subsequent clinical deterioration.

N-acetyl cysteine (NAC) is an attractive molecule for the proposed study because of two of its mechanistic properties. First, it is an established neuroprotective agent. NAC is a precursor to glutathione which is a primary detoxifier of reactive oxygen and other radical molecules which damage neuronal tissue (4-6). Glutathione deficiencies have been well documented in schizophrenia (7, 8). Second, NAC modulates glutamate release. NMDA hypofunction and altered glutamate release have been hypothesized to contribute to the cortical atrophy observed in early stage schizophrenia (9, 10). NAC has been shown to antagonize both the phencyclidine (PCP) effects of increased frontal glutamate levels and induction of social isolation in rodents (11). PCP is a pharmacological model of schizophrenia. In a controlled clinical trial of patients with chronic schizophrenia, NAC improved mismatch negativity, a pre-attentive measure of cortical information processing that has been consistently implicated in the pathophysiology of schizophrenia and has been shown to correlate with cortical erosion in early stage patients (12, 13). In a double-blind, placebo controlled clinical trial of chronic schizophrenic patients, NAC significantly improved general psychopathology scores, negative symptoms and extrapyramidal symptoms (14). NAC was well tolerated with no significant effects on any safety parameter or adverse events. The favorable tolerability of NAC has been further demonstrated in a recent study conducted at IUSM Riley Hospital in children (ages 4 to 12 years) with autism at relatively high doses (dose range of 900 to 4200 mg/day) in which there were no serious adverse events reported and NAC was well tolerated (15).

The investigators propose to determine if NAC has disease modifying potential in early stage schizophrenia. The investigators hypothesize that NAC will improve measures of cortical integrity in early stage schizophrenia and these brain effects will be related to improvements in negative symptoms and cognitive functioning. Primary outcome measures in the trials will be serial assessments of cortical integrity using magnetic resonance structural (cortical thickness, cortical volume, diffuses tensor imaging, DTI). In addition the investigators will assess the possible effects of NAC treatment on other parameters linked to cortical erosion including fMRI coupled with working memory and semantic memory tasks, MR spectroscopy (cortical glutathione, N-acetylaspartate, and glutamine/glutamate levels) and electrophysiological measures (e.g., mismatch negativity, P300). The investigators will also determine the relationship between effects of NAC on negative symptoms, positive symptoms, functional status, cognition (BACS), and safety parameters; and brain indices.

ELIGIBILITY:
SUBJECTS DIAGNOSED WITH A PSYCHOTIC DISORDER

Inclusion Criteria:

* Patients with a DSM-IV diagnosis of schizophrenia, schizophreniform, schizoaffective, psychosis disorder NOS
* Age range 16-35 years
* Male or female
* Within 2 years of the first onset of psychotic symptoms that resulted in work/school/social dysfunction and/or treatment (PI will review potential subjects who have been experiencing symptoms >2 years but <5 years and will allow to enter the trial on a case-by-case basis)
* Ability to provide informed consent and/or assent (all subjects)
* For subjects 16 and 17 years of age, parental/guardian consent

Exclusion Criteria:

* Unstable medical conditions
* Active seizure disorder
* Pregnant or lactating women
* Females unwilling to utilize birth control
* Implanted pacemaker, medication pump, vagal stimulator, deep brain stimulator, TENS unit, or ventriculoperitoneal shunt (because of MR studies).
* Known IQ less than 70
* DSM-IV-TR diagnosis of substance dependence (with the exception of nicotine or caffeine dependence)
* Psychotic symptoms secondary to substance use
* Considered a high risk for suicidal acts - active suicidal ideation with intent to act as determined by clinical interview

HEALTHY CONTROL SUBJECTS

The comparison subjects will consist of 40 healthy normal volunteers recruited from the community who will be age and gender matched to subjects diagnosed with a psychotic disorder entering the NAC treatment study

Inclusion Criteria:

1. Age range of 18-30 (inclusive) and able to give voluntary informed consent (Note: Subjects diagnosed with a psychotic disorder under the age of 18 will be age matched to control subjects aged 18).
2. Male or Female

Exclusion Criteria:

1. Current severe mental disorder (Schizophrenia, schizophreniform disorder, other psychotic disorders, bipolar disorder, major depressive disorder)
2. Known/documented IQ < 70
3. Pregnant or lactating women
4. Acute, serious, or unstable medical condition
5. Metallic implants or other contraindication to MRI (including but not limited to: Implanted pacemaker, medication pump, vagal stimulator, deep brain stimulator, TENS unit, or ventriculoperitoneal shunt)
6. First degree relative with a psychotic disorder (i.e. schizophrenia, schizophreniform, schizoaffective, psychosis disorder NOS, substance induced psychosis, major depression with psychotic features, or bipolar disorder with psychotic features).
7. Current DSM-IV-TR diagnosis of substance abuse or dependence (with the exception of nicotine or caffeine) as diagnosed within the 6 months prior to screening visit
8. Known history of seizure disorder, head trauma, stroke, traumatic brain injury, significant loss of consciousness

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2011-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Prevention and Recovery Center for Early Psychosis (PARC), Indianapolis, Indiana
  - Indiana University Psychotic Disorders Clinic, Indianapolis, Indiana

REFERENCES:
- [Derived] Breier A, Liffick E, Hummer TA, Vohs JL, Yang Z, Mehdiyoun NF, Visco AC, Metzler E, Zhang Y, Francis MM. Effects of 12-month, double-blind N-acetyl cysteine on symptoms, cognition and brain morphology in early phase schizophrenia spectrum disorders. Schizophr Res. 2018 Sep;199:395-402. doi: 10.1016/j.schres.2018.03.012. Epub 2018 Mar 24. PMID 29588126

RESULTS

PARTICIPANT FLOW:
Groups:
- N-Acetyl Cysteine: NAC and matched placebo will be supplied in unmarked capsules. Each NAC capsule will contain 600 mg of NAC. Dosing will begin at 600 mg/d and titrated up over 5 weeks until a maximum dose of 3600 mg/d is reached. Dose adjustments downward to 1920 mg/d will be permitted if tolerability issues are encountered at the maximum dose.
Period: Overall Study
Arm/Group | N-Acetyl Cysteine | Sugar Pill
Started | 30 | 30
Completed | 14 | 18
Not Completed | 16 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | N-Acetyl Cysteine | Sugar Pill | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 3
  Between 18 and 65 years | 28 | 29 | 57
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.2 (4.2) | 25.0 (5.2) | 23.1 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 23 | 24 | 47
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Cortical Thickness
Description: We anticipate that 12 months treatment with NAC as an add-on treatment will show significantly less cortical erosion as measured by cortical thickness than treatment with placebo
Time Frame: 12 months
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | N-Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 30 | 30
mm
  Left Total Cortical Thickness at 52 Weeks | 2.53 (0.03) | 2.54 (0.03)
  Right Total Cortical Thickness at 52 weeks | 2.51 (0.03) | 2.52 (0.03)
  Left Caudal Middle Frontal Thickness at 52 Weeks | 2.59 (0.04) | 2.57 (0.04)
  Right Caudal Middle Frontal Thickness at 52 Weeks | 2.49 (0.04) | 2.49 (0.05)
  Left Middle Temporal Thickness at 52 Weeks | 2.84 (0.04) | 2.87 (0.05)
  Right Middle Temporal Thickness at 52 Weeks | 2.91 (0.04) | 2.95 (0.05)
  Left Superior Parietal Thickness at 52 Weeks | 2.16 (0.03) | 2.21 (0.04)
  Right Superior Parietal Thickness at 52 Weeks | 2.17 (0.03) | 2.18 (0.04)

2. Secondary Outcome: Working Memory
Description: determine if 12 months of NAC add-on treatment is superior to placebo as determined by brain activity during n-back working memory task during fMRI.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: Bold signal change
Arm/Group | N-Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 30 | 30
Bold signal change
  Baseline pre exposure to NAC | 0.299 (.20) | 0.356 (.24)
  6 months exposure to NAC | 0.351 (.24) | 0.398 (.28)
  12 months exposure to NAC | 0.315 (.185) | 0.406 (.23)

3. Secondary Outcome: Number of Participants With Glutamine/Glutamate Level Changes
Description: Identify number of participants with 12 months of NAC treatment who had glutamine/glutamate level changes as measured by cortical magnetic resonance spectroscopy measures.
Time Frame: 12 months
Population: Several subjects were excluded from the MR spectroscopy measures due to visible motion between image acquisitions. Data were not collected for the Placebo group.
Measure: Count of Participants; unit: Participants
Groups:
- NAC Treated Early Psychosis Patients: Longitudinal concentrations of glutamine/glutamate (Glx) levels across three scans for NAC treated patients
Arm/Group | NAC Treated Early Psychosis Patients | Placebo Group
Number analyzed (Participants) | 18 | 0
Participants | 18 | 0
Statistical Analysis 1: Comparison: NAC Treated Early Psychosis Patients; Test type: Superiority; p = 0.32, ANOVA

4. Secondary Outcome: Attention Measures
Description: determine if 12 months of NAC add-on treatment is superior to placebo for attention measures (e.g., mismatch negativity, P300) as measured by electrophysiology methods. Electrophysiology measures will be recorded from a 64 channel, silver/silver-chloride scalp electrode montage.
Time Frame: 12 months
Measure: Least Squares Mean (Standard Error); unit: Hz
Arm/Group | N-Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 30 | 30
Hz
  EEG Alpha power | 3.81 (0.40) | 4.18 (0.73)
  EEG Delta power | 2.96 (0.25) | 3.46 (0.35)
  EEG Gamma power | 0.37 (0.03) | 0.47 (0.05)
  EEG Theta power | 1.33 (0.30) | 1.33 (0.35)
  Auditory Steady State Response 40 Hz | 0.05 (0.01) | 0.06 (0.01)

5. Secondary Outcome: Symptoms of a Psychotic Disorder
Description: Determine if 12 months of NAC add-on treatment is superior to placebo for symptom management of a psychotic disorder as assessed by the Positive and Negative Syndrome Scale (PANSS). The PANSS is a semi-structured interview, containing 30 items that assess positive, negative, and general psychopathology symptoms. Positive symptoms=7 items, negative symptoms=7 items, and general psych.=16 items. Scores for each item range from 1-absent to 7-extreme. To calculate total score, all items on the scale are summed to yield a score from 30-210,a lower score reflecting fewer symptoms. To calculate factor scores various items from positive, negative, and general psych. are summed together to yield Cognitive/Disorganized, Negative, and Positive factor scores. Cog/Disorg factor scores sum 7 items, ranging from 7-49. Neg factor scores sum 7 items, ranging from 7-49. Pos factor scores sum 8 items, ranging from 8-56. For all factor scores a lower score reflects less symptom severity.
Time Frame: 12 months
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | N-Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 30 | 30
scores on a scale
  PANSS Total Score at 52 Weeks | 46.79 (2.24) | 56.44 (2.32)
  PANSS Cognitive/Disorganized Factor at 52 Weeks | 11.09 (0.68) | 13.68 (0.70)
  PANSS Negative Symptom Factor at 52 Weeks | 10.35 (1.02) | 13.22 (1.06)
  PANSS Positive Symptom Factor at 52 Weeks | 14.77 (1.05) | 16.38 (1.09)

6. Secondary Outcome: Cognitive Functioning
Description: determine if 12 months of NAC add-on treatment is superior to placebo for cognitive functioning as measured by the Brief Assessment of Cognition in Schizophrenia (BACS). The BACS is a battery specifically designed to measure treatment-related changes in cognition by utilizing 6 tasks, and has alternate forms, thus minimizing practice effects. Each task generates a raw score (with a higher score indicating better performance): verbal memory 0-75; digit sequencing 0-28; token motor task 0-100; semantic&letter fluency 0-148; symbol coding 0-110; and tower of London 0-22. The raw scores are used to generate a composite score that is calculated by summing t-scores derived by comparisons with a normative sample of 404 healthy controls. The six brief assessments' t-scores, are summed, and averaged to provide a composite t-score. The composite score min and max are between -43 and 100. A higher score indicating better cognitive performance.
Time Frame: Baseline and 12 months
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | N-Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 30 | 30
scores on a scale
  BACS Composite Score Baseline | 26.91 (3.22) | 27.70 (3.35)
  BACS Composite Score at 52 Weeks | 30.03 (3.22) | 29.37 (3.36)

7. Secondary Outcome: Functional Status
Description: determine if 12 months of NAC add-on treatment is superior to placebo for functional measures as measured by the Personal and Social Performance Scale (PSP). The PSP scale is a 100-point, single item, clinician rated scale to assess 4 domains of functioning, including personal and social relationships, socially useful activities, self care and disturbing and aggressive behaviors. A score from 0-100 is generated, with a higher score representing better performance.
Time Frame: Baseline and 12 months
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | N-Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 30 | 30
scores on a scale
  PSP Adjusted Score at Baseline | 62.51 (2.26) | 64.46 (2.35)
  PSP Adjusted Score at 52 Weeks | 64.51 (2.33) | 65.44 (2.42)

8. Secondary Outcome: Mismatch Negativity Voltage Differences
Description: Determine if 12 months of NAC add-on treatment is superior to placebo for attention measures as measured by the voltage of the Mismatch Negativity (MMN) of the event-related potential. The voltage of the peak MMN response was measured at the Fz electrode site.
Time Frame: 12 months
Measure: Least Squares Mean (Standard Error); unit: microvolts
Arm/Group | N-Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 30 | 30
microvolts | -2.51 (0.28) | -3.44 (0.38)

9. Primary Outcome: Cortical Volume
Description: We anticipate that 12 months treatment with NAC as an add-on treatment will show a difference in cortical volume than treatment with placebo
Time Frame: 12 months
Measure: Least Squares Mean (Standard Error); unit: mm^3
Arm/Group | N-Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 30 | 30
mm^3
  Total Cortical Gray Matter Volume at 52 Weeks | 233.0 (5.2) | 235.8 (6.0)
  Total Cortical White Matter Volume at 52 Weeks | 423.8 (11.5) | 418.5 (13.1)

10. Secondary Outcome: Symptoms of a Psychotic Disorder
Description: determine if 12 months of NAC add-on treatment is superior to placebo for symptom management of a psychotic disorder as assessed by the Clinical Global Impressions Severity Scale (CGI-S). The CGI-S is used for repeated evaluations of global psychopathology and is a 7 point Likert scale rating severity on a scale of 1 (normal, not ill) to 7 (very severely ill).
Time Frame: 12 months
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | N-Acetyl Cysteine | Sugar Pill
Number analyzed (Participants) | 30 | 30
scores on a scale | 2.78 (0.18) | 3.00 (0.19)

ADVERSE EVENTS:
Arm/Group | N-Acetyl Cysteine | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 3/30 | 2/30
Other Adverse Events (participants affected / at risk) | 28/30 | 27/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-Acetyl Cysteine (N=30) | Sugar Pill (N=30)
Asthma Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Psychosis Exacerbation (Psychiatric disorders) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-Acetyl Cysteine (N=30) | Sugar Pill (N=30)
Headache (Nervous system disorders) | 3 (3) | 2 (2)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 2 (2)
Sedation (General disorders) | 2 (2) | 3 (3)
Insomnia (General disorders) | 3 (3) | 2 (2)
Illness Exacerbation (Psychiatric disorders) | 3 (3) | 0 (0)
Depressed Mood (Psychiatric disorders) | 4 (4) | 4 (5)
Dyskinesia (Nervous system disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Nausea and Vomiting (Gastrointestinal disorders) | 3 (3) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 0 (0)
Nasal Congestion (General disorders) | 1 (1) | 2 (2)
Toothache (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 2 (2) | 3 (3)
Weight Gain (Metabolism and nutrition disorders) | 3 (3) | 6 (6)
Hyperlipidemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Dyspepsia (Cardiac disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No